CLINICAL TRIAL: NCT04833218
Title: Propranolol Versus Propranolol and Clonidine in Sympathetic Hyperactivity After Moderate Traumatic Brain Injury
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Fatma Rabea Mohammed, assistant lecturer, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 389:1/2020
Record Dates: First submitted 2021-03-10; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-01

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Propranolol; Clonidine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- propranolol group (Active Comparator): we will give propranolol 40 milligram tablet twice daily in orogastric or nasogastric tube
  Interventions: Drug: Propranolol
- propranolol clonidine (Active Comparator): we will give propranolol 20 milligram tablet twice daily and clonidine 150 microgram tablet twice daily in orogatric or nasogastric tube
  Interventions: Drug: Propranolol
- control group (No Intervention): we will give conventional treatment, no propranolol nor clonidine

INTERVENTIONS:
Drug: Propranolol — Test of catecholamines level in moderate traumatic brain injury
  Other Names: Clonidine
  Arms: propranolol clonidine; propranolol group

SUMMARY:
evaluation of the effect of Propranolol versus propranolol and clonidine on decreasing sympathetic hyperactivity after moderate traumatic brain injury

DETAILED DESCRIPTION:
measuring catecholamine levels after moderate traumatic brain injury after giving propranolol and clonidine

ELIGIBILITY:
Inclusion Criteria:

* GCS on admission between 9 and 12 age 18 up to 60 years both sexes

Exclusion Criteria:

* history of heart disease, cardiac arrhythmia and myocardial infarction diagnosis ofpreexisting brain dysfunction. impending brain herniation and craniotomy diagnosis of spinal cord injuries. diagnisis of severe liver and renal disease current use of beta blocker and or alpha agonist current using of intravenous vasopressor contraindication to enteral feeding and can not swallow pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-01-31 (Actual); Primary Completion 2021-06-22 (Estimated); Study Completion 2021-07-22 (Estimated)

PRIMARY OUTCOMES:
catecholamine level on day 7 | seven days
  measuring catecholamine level on day 7 after giving study drugs

SECONDARY OUTCOMES:
mean arterial blood pressure every 4 hours herat rate every 4 hours temperature every 4 hours respiratory rate every 4 hours | 7 days
  measuring hemodynamics every 4 hours
Glascow coma scale | 7 days
  measuring glascow coma scale twice daily between 9 and 12 and higher score means better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Amany Khairy, MD, Study Chair — Professor
Locations (1):
- Faculty Of Medicine, Minya, Egypt